CLINICAL TRIAL: NCT01068834
Title: Additional KIF6 Risk Offers Better Adherence to Statins
Acronym: AKROBATS
Status: Completed | Type: Observational
Sponsor: Medco Health Solutions, Inc. (Industry)
Collaborators: Celera Genomics (Industry)
Responsible Party: Scott L Charland, Pharm.D. Director, Clinical Research & Health Outcomes, Personalized Medicine, Medco Health Solutions, Inc
Other Study IDs: AKROBATS
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Diseases; Dyslipidemia
Keywords: Adherence; Statins; Kinesin-like protein 6
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- KIF6 tested: Recruited subjects, completing a valid KIF6 test with results
  Interventions: Genetic: KIF6 genetic test
- KIF6 test naïve: Database matched cohort not receiving a KIF6 test

INTERVENTIONS:
Genetic: KIF6 genetic test — KIF6 carrier status with interpretation sheet provided to subject
  Groups: KIF6 tested

SUMMARY:
Many patients prescribed statins to lower their cholesterol stop taking their statin over time. The purpose of this study is to determine whether providing subjects their KIF6 carrier status (associated with increased cardiovascular event risk) will improve adherence to statin medications.

DETAILED DESCRIPTION:
Coronary Heart Disease (CHD) remains a significant problem in the US, causing about 1 of every 5 deaths in 2005. In 2009, approximately 1.3 million Americans will have a new/recurrent myocardial infarction. Coronary heart disease (CHD) includes myocardial infarction, stable or unstable angina, demonstrated myocardial ischemia detected by noninvasive testing, and a history of coronary artery procedures (such a stent or bypass). Currently, "statins" are recommended by the AHA to manage elevated low-density lipoprotein-cholesterol (LDL-C). Unfortunately, the discontinuation of statins is quite substantial. For example, a large cohort study of older patients found that 2-year statin adherence rates were approximately 40% for acute coronary syndrome patients, 36% for chronic coronary artery disease, and 25% for primary prevention and is associated with increased mortality, hospitalizations, and costs. Recently, the kinesin 6 (KIF6) gene has been associated with a 30-55% increase in cardiovascular events in individuals carrying one or two risk variants (~57% of the white population) in multiple prospective studies. Furthermore, KIF6 carriers receiving a "statin" have a substantial greater cardiovascular risk reduction (-34 to 50%) when using a "statin" compared to those that are non-carriers using a statin (6 to 20%). In this prospective, open label, trial, recruited subjects recently started on statin therapy will be provided information about their KIF6 carrier status and followed for 6 months to determine their "statin" adherence. Additionally, quality of life and factors adherence will be measured at baseline and after 6 months. Finally, pharmacy records will be evaluated for up to 1-year to determine statin discontinuation rates.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age
* New statin prescription
* Medco RationalMed® Program
* Data contains patient contact information (e.g. phone number)
* Data contains provider contact information
* Willing to sign informed consent and send KIF6 test results to their provider

Exclusion Criteria:

* Statin prescription in the previous 6 months
* Subject refusal to participate in this study (record reason from subject)
* Physician refusal to participate in this study (record reason from provider)
* Anticipated statin discontinuation within 6 months
* Any condition that would prevent the subject from completing the 6 month study follow-up period
* Subject with "no contact red flag"
* Subject residing in NY, NJ, MA, PA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (> 18y/o) newly started on either a brand name or generic statin (atorvastatin, fluvastatin, lovastatin, pitavastatin, pravastatin, rosuvastatin, and simvastatin with or without ezetimibe) being followed in Medco's RationalMed® program
Sampling Method: Non-Probability Sample
Enrollment: 1282 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Proportion of days covered with statins in subjects tested for KIF6 status compared to statin-treated subjects who are not offered the test (KIF6 test naïve) | 6 months

SECONDARY OUTCOMES:
To evaluate characteristics of subjects who agree to be tested for KIF6 carrier status | 6 months
To evaluate adherence rate or medication gap in KIF6 carriers compared to KIF6 test naïve | 6 months
To compare the PDC, MPR and or gap in KIF6 carriers and KIF6 non-carriers | 6 months
To compare statin discontinuation rates between KIF6 carriers, non-carriers, and KIF6 test naïve subjects | up to 12 months
Shift in PDC between non-adherent, partially adherent, and adherent (< 0.2, >0.2 to <0.8, > 0.8, respectively) between KIF6 tested and KIF6 test naïve subjects | 6 month
To compare SF-12 v2 summary measure scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS); and, a health utility index (SF-6D.), as well as, the Morisky Adherence Scale between KIF6 carriers and non-carriers | 6 months
To determine cardiovascular costs associated with PDC | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Charland, PharmD, Principal Investigator — Medco Health Solutions, Inc.; James J Devlin, PhD, Principal Investigator — Celera Genomics
Locations (1):
- Medco Health Solutions, Inc, Franklin Lakes, New Jersey, United States

REFERENCES:
- [Background] Lloyd-Jones D, Adams R, Carnethon M, De Simone G, Ferguson TB, Flegal K, Ford E, Furie K, Go A, Greenlund K, Haase N, Hailpern S, Ho M, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott M, Meigs J, Mozaffarian D, Nichol G, O'Donnell C, Roger V, Rosamond W, Sacco R, Sorlie P, Stafford R, Steinberger J, Thom T, Wasserthiel-Smoller S, Wong N, Wylie-Rosett J, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2009 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2009 Jan 27;119(3):e21-181. doi: 10.1161/CIRCULATIONAHA.108.191261. Epub 2008 Dec 15. No abstract available. PMID 19075105
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Jackevicius CA, Mamdani M, Tu JV. Adherence with statin therapy in elderly patients with and without acute coronary syndromes. JAMA. 2002 Jul 24-31;288(4):462-7. doi: 10.1001/jama.288.4.462. PMID 12132976
- [Background] Ho PM, Magid DJ, Shetterly SM, Olson KL, Maddox TM, Peterson PN, Masoudi FA, Rumsfeld JS. Medication nonadherence is associated with a broad range of adverse outcomes in patients with coronary artery disease. Am Heart J. 2008 Apr;155(4):772-9. doi: 10.1016/j.ahj.2007.12.011. PMID 18371492
- [Background] Iakoubova OA, Sabatine MS, Rowland CM, Tong CH, Catanese JJ, Ranade K, Simonsen KL, Kirchgessner TG, Cannon CP, Devlin JJ, Braunwald E. Polymorphism in KIF6 gene and benefit from statins after acute coronary syndromes: results from the PROVE IT-TIMI 22 study. J Am Coll Cardiol. 2008 Jan 29;51(4):449-55. doi: 10.1016/j.jacc.2007.10.017. PMID 18222355
- [Background] Iakoubova OA, Tong CH, Rowland CM, Kirchgessner TG, Young BA, Arellano AR, Shiffman D, Sabatine MS, Campos H, Packard CJ, Pfeffer MA, White TJ, Braunwald E, Shepherd J, Devlin JJ, Sacks FM. Association of the Trp719Arg polymorphism in kinesin-like protein 6 with myocardial infarction and coronary heart disease in 2 prospective trials: the CARE and WOSCOPS trials. J Am Coll Cardiol. 2008 Jan 29;51(4):435-43. doi: 10.1016/j.jacc.2007.05.057. PMID 18222353
- [Background] Morrison AC, Bare LA, Chambless LE, Ellis SG, Malloy M, Kane JP, Pankow JS, Devlin JJ, Willerson JT, Boerwinkle E. Prediction of coronary heart disease risk using a genetic risk score: the Atherosclerosis Risk in Communities Study. Am J Epidemiol. 2007 Jul 1;166(1):28-35. doi: 10.1093/aje/kwm060. Epub 2007 Apr 18. PMID 17443022
- [Background] Shiffman D, Chasman DI, Zee RY, Iakoubova OA, Louie JZ, Devlin JJ, Ridker PM. A kinesin family member 6 variant is associated with coronary heart disease in the Women's Health Study. J Am Coll Cardiol. 2008 Jan 29;51(4):444-8. doi: 10.1016/j.jacc.2007.09.044. PMID 18222354
- [Background] Shiffman D, O'Meara ES, Bare LA, Rowland CM, Louie JZ, Arellano AR, Lumley T, Rice K, Iakoubova O, Luke MM, Young BA, Malloy MJ, Kane JP, Ellis SG, Tracy RP, Devlin JJ, Psaty BM. Association of gene variants with incident myocardial infarction in the Cardiovascular Health Study. Arterioscler Thromb Vasc Biol. 2008 Jan;28(1):173-9. doi: 10.1161/ATVBAHA.107.153981. Epub 2007 Nov 1. PMID 17975119